CLINICAL TRIAL: NCT00115323
Title: Individualized Interventions to Improve Asthma Adherence
Brief Title: Comparison of Two Medication Adherence Strategies to Improve Asthma Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andrea Apter, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190; R01HL073932 (NIH)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Problem solving intervention
  Interventions: Behavioral: Problem Solving
- 2 (Active Comparator): Attention control intervention
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Problem Solving — Problem solving intervention
  Arms: 1
Behavioral: Attention Control — Attention control intervention
  Arms: 2

SUMMARY:
This is a randomized, controlled study that will compare two medication adherence strategies in adults with moderate or severe persistent asthma as a method for improving or maintaining treatment adherence.

DETAILED DESCRIPTION:
Low-income minority adults have excessively high rates of morbidity from asthma. Poor medication adherence has been documented in these individuals and contributes to the high morbidity level. This study will compare a Problem Solving intervention with an Attention Control intervention to improve and sustain asthma self-management in a clinical setting. This study will include strategies to address contextual factors related to adherence. Participants will be recruited from clinics that serve minority and low-income individuals.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment for asthma at one of the participating clinics
* Moderate or severe persistent asthma according to the NHLBI Guidelines
* Current use of prescribed inhaled corticosteroids
* Evidence of reversible airflow obstruction, as indicated by the following two criteria:

  1. FEV1pp AND less than 80% at the time of study entry or within the 3 years prior to study entry
  2. An increase of greater than 15% and 200ml in FEV1 with asthma treatment over the last 3 years (if there is no record of such improvement, participants will be evaluated via spirometry pre- and post-bronchodilator at the first study visit. An increase in FEV1 or FVC greater than 12% and 200 ml in FEV1 30 minutes following albuterol administration will represent evidence of reversible airflow obstruction. If a spirometer is not immediately available, participants may be evaluated using a peak flow meter, which reports a PEF. A PEFpp less than 80% and an improvement of at least 60 L per minute after the administration of albuterol will represent evidence of reversible airflow obstruction)
* Has a functional telephone or mobile phone

Exclusion Criteria:

* Significant lung or cardiac disease (other than hypertension)
* Psychiatric illness, such as mania or schizophrenia, that may make it impossible to understand or carry out the Problem Solving intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2005-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed inhaled steroid regimen | Measured at Week 26

SECONDARY OUTCOMES:
FEV1 | Measured at Week 26
Quality of life factors | Measured at Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Apter, Study Chair — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Naimi DR, Freedman TG, Ginsburg KR, Bogen D, Rand CS, Apter AJ. Adolescents and asthma: why bother with our meds? J Allergy Clin Immunol. 2009 Jun;123(6):1335-41. doi: 10.1016/j.jaci.2009.02.022. Epub 2009 Apr 22. PMID 19395075
- [Background] Apter AJ, Garcia LA, Boyd RC, Wang X, Bogen DK, Ten Have T. Exposure to community violence is associated with asthma hospitalizations and emergency department visits. J Allergy Clin Immunol. 2010 Sep;126(3):552-7. doi: 10.1016/j.jaci.2010.07.014. PMID 20816190
- [Background] Apter AJ, Wang X, Bogen D, Bennett IM, Jennings RM, Garcia L, Sharpe T, Frazier C, Ten Have T. Linking numeracy and asthma-related quality of life. Patient Educ Couns. 2009 Jun;75(3):386-91. doi: 10.1016/j.pec.2009.01.003. Epub 2009 Feb 13. PMID 19217741
- [Background] Apter AJ, Cheng J, Small D, Bennett IM, Albert C, Fein DG, George M, Van Horne S. Asthma numeracy skill and health literacy. J Asthma. 2006 Nov;43(9):705-10. doi: 10.1080/02770900600925585. PMID 17092853
- [Background] Apter AJ, Paasche-Orlow MK, Remillard JT, Bennett IM, Ben-Joseph EP, Batista RM, Hyde J, Rudd RE. Numeracy and communication with patients: they are counting on us. J Gen Intern Med. 2008 Dec;23(12):2117-24. doi: 10.1007/s11606-008-0803-x. Epub 2008 Oct 2. PMID 18830764
- [Result] Apter AJ, Wang X, Bogen DK, Rand CS, McElligott S, Polsky D, Gonzalez R, Priolo C, Adam B, Geer S, Ten Have T. Problem solving to improve adherence and asthma outcomes in urban adults with moderate or severe asthma: a randomized controlled trial. J Allergy Clin Immunol. 2011 Sep;128(3):516-23.e1-5. doi: 10.1016/j.jaci.2011.05.010. Epub 2011 Jun 25. PMID 21704360